CLINICAL TRIAL: NCT00036569
Title: A Phase II Study of Pegylated Interferon Alfa-2b (Peg-Intron (TM)) in Children With Diffuse Pontine Gliomas
Brief Title: A Phase II Study of Pegylated Interferon Alfa 2b (PEG-Intron(Trademark)) in Children With Diffuse Pontine Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Katherine E. Warren, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020193; 02-C-0193; NCT00041145 (obsolete NCT alias)
Record Dates: First submitted 2002-05-10; First posted 2002-05-13 (Estimated); Results first posted 2012-02-13 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-01

CONDITIONS: Diffuse Intrinsic Pontine Glioma
Keywords: Brainstem Glioma; Pediatric; Interferon; MR Imaging; Angiogenesis; Brain Tumor; Glioma; Pediatric Brain Tumor
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Brain Neoplasms; Glioma | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interferon Alfa (Experimental): 0.3 mg/kg subcutaneously once a week for 4 weeks beginning 2-10 weeks after completion of radiation therapy and continued until disease progression or one of the other off study criteria.
  Interventions: Procedure: adjuvant therapy; Biological: pegylated interferon alfa

INTERVENTIONS:
Procedure: adjuvant therapy
Biological: pegylated interferon alfa — 0.3 mg/kg subcutaneously once a week for 4 weeks beginning 2-10 weeks after completion of radiation therapy and continued until disease progression or one of the other off study criteria.

SUMMARY:
Diffuse pontine gliomas are tumors on the pons portion of the brainstem. Their peak incidence is in children between 5 and 10 years old. Their location makes surgical resection impossible. Most patients are treated with radiation, which typically delays progression of the tumor for a median time of only about 6 months; median survival time is less than 1 year. The addition of chemotherapy has not improved the outcome.

Alpha, beta, and gamma interferons have been used to treat malignant brain tumors, with mixed results. Different doses and different methods of administration have been studied. Alpha interferon is usually given in high doses 2 or 3 times a week, but it has serious side effects at these doses. Recent studies have shown that administering chemotherapy more frequently at smaller doses (metronomic) may have a better effect against the tumor.

PEG-Intron(Trademark) is a form of interferon alpha combined with monomethoxy polyethylene glycol (PEG). It has a longer half-life than interferon alone, is administered once a week, and the long half-life reduces the peaks and troughs in blood levels.

This study will enroll 32 patients under age 21. The primary goals of the study are to determine if there is a difference in the 2-year survival rate of patients treated with radiation alone and those treated with radiation followed by PEG-Intron(Trademark) and to define the toxicities of PEG-Intron(Trademark) in the study doses. Secondary goals are to evaluate various magnetic resonance imaging (MRI) techniques for noninvasive monitoring of changes in the brainstem and to evaluate neuropsychological function.

In this study, PEG-Intron(Trademark) will be administered subcutaneously once a week at low doses (0.3 microgram per kilogram of body weight) for a 4-week cycle. The cycles will be repeated indefinitely until progression of disease or serious side effects develop. For less severe effects, the dose will be lowered and the patient may remain in the study. For more severe effects, the dose will be discontinued. Patients in the study may receive supportive medication but may not receive other forms of chemotherapy.

Patients or their caregivers will be instructed in how to inject the drug. Patients and/or caregivers will be asked to maintain a diary documenting the dose, site of administration, and any side effects. The diary will be reviewed at each National Cancer Institute (NCI) visit. Patients will return to NCI before cycles 2 and 3. If there are no significant side effects, patients may then return to NCI before every other cycle, indefinitely (i.e., before cycles 5, 7, 9, etc.).

Patients will undergo the following tests and procedures:

* Physical examination, including neurologic exam, monthly
* Complete blood count, differential, and platelet count weekly during cycle 1 and every 2 weeks thereafter if no severe side effects occur
* Blood chemistries weekly during cycle 1 and every 2 weeks thereafter if no severe side effects occur
* Endocrine function tests before each cycle
* Urinalysis before each cycle
* MRI of the brain before cycles 1, 2, 3, 5, 7, and every other month; patients may also have proton magnetic spectroscopic imaging performed at the time of the MRI

DETAILED DESCRIPTION:
Background:

Children with diffuse pontine gliomas have a dismal prognosis. Because surgery in this area is difficult, radiation therapy has been the mainstay of treatment. Although some children may improve clinically after radiation therapy, the effect is short-lived and almost all progress within several months. Chemotherapy has not had a significant impact on survival. Interferon-alpha is a cytokine that has been studied in patients with gliomas and has demonstrated some activity in prior clinical trials.

Objectives:

* To compare the 2-year survival of pediatric patients with diffuse pontine gliomas receiving weekly subcutaneous low-dose pegylated interferon alfa-2b (PEG-Intron[TM]) injections after standard radiation therapy versus historical controls who have received radiation therapy alone.
* To define the toxicities of weekly low-dose pegylated interferon alfa-2b (PEG-Intron(Trademark)) in pediatric patients.

Eligibility:

Age: Patients must be less than or equal to 21 years of age.

Histological Diagnosis: Histologic confirmation is not required for this study. Patients must have a diffuse pontine glioma as diagnosed by MRI criteria below.

Radiologic Appearance: Patients must have a diffuse intrinsic tumor with the epicenter presumed to be in the pons. The T-2 weighted sequence must reveal a diffuse signal abnormality involving at least 50 percent of the pons.

Prior Therapy: The patient must have received adequate radiation therapy. Radiation must be completed between 2-10 weeks prior to the start of treatment with Peg-Intron[TM].

Design:

In this study, we plan to administer pegylated interferon alfa-2b (PEG-Intron[TM]) subcutaneously once a week to pediatric patients with diffuse pontine gliomas who have completed radiation therapy. The endpoint of the trial will be 2-year survival compared to historical controls.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age: Patients must be less than or equal to 21 years of age.

Histological diagnosis: Histologic confirmation is not required for this study. Patients must have a diffuse pontine glioma as diagnosed by magnetic resonance imaging (MRI) criteria below.

Radiographic Appearance: Patients must have a diffuse intrinsic tumor with the epicenter presumed to be in the pons. The T-2 weighted sequence must reveal a diffuse signal abnormality involving at least 50 percent of the pons.

Prior therapy: The patient must have received adequate radiation therapy. (Radiation must be completed between 2-10 weeks prior to the start of treatment with Peg-Intron (TM).

Performance status: Patients should have an Cooperative Oncology Group (ECOG) performance status of 0, 1, 2, or 3 (see below). Patients who are unable to walk because of paralysis, but who are up in a wheel chair will be considered ambulatory for the purpose of calculating the performance score.

ECOG Performance Status:

Score--Clinical Status

0--Asymptomatic

1. -Symptomatic, fully ambulatory
2. -Symptomatic, in bed less than 50 percent of the day
3. -Symptomatic, in bed greater than 50 percent of the day but not bedridden
4. -Bedridden

   Hematological function: Patients must have adequate bone marrow function defined as a peripheral absolute granulocyte count of greater than 1000/mm^3, hemoglobin greater than 8 gm/dL, and platelet count greater than 100,000/mm^3. Patients may be transfused with red blood cells (RBC's) or platelets to achieve these parameters.

   Hepatic function: Patients must have adequate liver function, defined as total bilirubin less than 2.5 times the upper limit of normal, direct bilirubin within normal limits, and serum glutamic pyruvic transaminase (SGPT) less than 2.0 times the upper limit of normal. Patients with Gilbert Syndrome are excluded from both the total and direct bilirubin requirements. (Gilbert Syndrome is found in 3-10 percent of the general population and is characterized by mild, chronic hyperbilirubinemia in the absence of liver disease or overt hemolysis.)

   Renal function: Patients must have an age-adjusted normal serum creatinine (see below) OR a creatinine clearance greater than or equal to 60 mL/min/1.73 m^2.

   Age (Years)---Maximum Serum Creatinine (mg/dl)

   less than or equal to 5---0.8

   greater than 5 and less than or equal to 10---1.0

   greater than 10 less than or equal to 15---1.2

   greater than 15---1.5

   Steroids: Patients on steroids must be on a stable or decreasing dose of steroids for greater than or equal to 1 week prior to study entry.

   Informed consent: All patients or their legal guardians (if the patient is less than 18 years old) or DPA must sign a document of informed consent indicating their understanding of the investigational nature and the risks of this study. When appropriate, pediatric patients will be included in all discussions in order to obtain verbal assent.

   Durable Power of Attorney (DPA): Assignment of DPA to a family member or guardian should be offered to all patients 18 to 21 years of age.

   EXCLUSION CRITERIA:

   Patients with known or suspected neurofibromatosis-1

   Patients who have received prior chemotherapy, including radiosensitizers, or who are currently receiving other investigational chemotherapeutic agents

   Patients with a known hypersensitivity to interferon-alpha

   Pregnant or breast-feeding females are excluded because the effects of pegylated interferon alfa-2b (PEG-Intron (TM)) on the unborn fetus are unknown.

   Patients with clinically significant unrelated systemic illness (including autoimmune disease, serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) which in the judgment of the Principal or Associate Investigators would compromise the patient's ability to tolerate this therapy or are likely to interfere with the study procedures or results.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2002-05; Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Warren, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Packer RJ, Nicholson HS, Vezina LG, Johnson DL. Brainstem gliomas. Neurosurg Clin N Am. 1992 Oct;3(4):863-79. PMID 1392581
- [Background] Freeman CR, Farmer JP. Pediatric brain stem gliomas: a review. Int J Radiat Oncol Biol Phys. 1998 Jan 15;40(2):265-71. doi: 10.1016/s0360-3016(97)00572-5. PMID 9457808
- [Background] Barkovich AJ, Krischer J, Kun LE, Packer R, Zimmerman RA, Freeman CR, Wara WM, Albright L, Allen JC, Hoffman HJ. Brain stem gliomas: a classification system based on magnetic resonance imaging. Pediatr Neurosurg. 1990-1991;16(2):73-83. doi: 10.1159/000120511. PMID 2132928
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-C-0193.html
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug information — http://druginfo.nlm.nih.gov/drugportal/drugportal/jsp
- See also: United States FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interferon Alfa
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Interferon Alfa
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 6.28 (3.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 13
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
  Black | 4
  Asian or Pacific Islander | 2
  Native Hawaiian | 1
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Two Year Survival of Pediatric Patients With Diffuse Pontine Gliomas
Description: Survival is measured from the date the patient is registered onto the protocol until the day of death and the date of diagnosis to the date of patient death.
Time Frame: 8 yrs 6 mo 0 days
Measure: Number; unit: Percentage of patients
Arm/Group | Interferon Alfa
Number analyzed (Participants) | 32
Percentage of patients | 14.29

2. Secondary Outcome: Median Time to Progression
Description: Time between the final day of treatment to the day of disease progression.
Time Frame: 8 yrs 11 mo 22 days
Measure: Number; unit: Days
Arm/Group | Interferon Alfa
Number analyzed (Participants) | 32
Days | 235

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 8 yrs 11 mo 22 days
Measure: Number; unit: Participants
Arm/Group | Interferon Alfa
Number analyzed (Participants) | 32
Participants | 32

4. Secondary Outcome: Mean Quality of Life (QOL) Score at Baseline and Follow-Up
Description: QOL questionnaires will be performed prior to every cycle for patients age 6-18 years and their parents until cycle 27 and then prior to every third cycle until cycle 52 when the evaluations will become annual. The QOL (NIH Impact of Pediatric Illness Scale) is too detailed to be described and/or shown here. It is a questionnaire made up of approximately 40 questions-the answers are ranked from 1 to 5 with 5 being no impact and 1 being significant impact-For further details see the protocol.
Time Frame: once a week for 4 weeks beginning 2-10 weeks after completion of radiation therapy and continued until disease progression or one of the other off study criteria.
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- QOL Score at Baseline; QOL Score at Follow-up: 0.3 mg/kg subcutaneously once a week for 4 weeks beginning 2-10 weeks after completion of radiation therapy and continued until disease progression or one of the other off study criteria.
Arm/Group | QOL Score at Baseline | QOL Score at Follow-up
Number analyzed (Participants) | 11 | 11
Units on a scale | 3.59 (0.11) [3.59, to 3.89,] | 3.89 (0.11)

5. Secondary Outcome: Number of Participants With a Metabolic and Biological Change in the Brainstem Through Magnetic Resonance Imaging (MRI) Techniques
Description: MRI of the brain will be performed at the NCI prior to cycles 1, 2, 3, 5, 7, and continuing every other month until cycle 27. Following cycle 27 the patient will have an MRI performed every third cycle until cycle 52 at which time they will have an MRI performed annually, and when clinically indicated. Baseline MR images are compared with MR images performed during the various cycles (e.g. cycles 1, 2, 3...) Imaging was exploratory and the degree of change that is considered clinically significant rather than technique related is still being explored.
Time Frame: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Interferon Alfa
Number analyzed (Participants) | 32
Participants | 32

ADVERSE EVENTS:
Arm/Group | Interferon Alfa
Serious Adverse Events (participants affected / at risk) | 32/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Alfa (N=32)
ALT (Investigations) | 7 (8)
Ataxia (Nervous system disorders) | 1 (1)
Diplopia (Eye disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Leukopenia (Investigations) | 9 (16)
Lymphopenia (Investigations) | 9 (20)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy-cranial (Nervous system disorders) | 12 (42)
Neuropathy-motor (Nervous system disorders) | 3 (3)
Neutropenia (Investigations) | 12 (32)
Pyramidal tract dysfunction (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Alfa (N=32)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase (ALT) (Investigations) | 12 (24)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase (AST) (Investigations) | 7 (17)
Ataxia (Nervous system disorders) | 0 (0)
Bilirubin (Investigations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 3 (4)
Diplopia (Eye disorders) | 0 (0)
Fatigue (General disorders) | 3 (4)
Fever (General disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (4)
Hemoglobin (Investigations) | 6 (26)
Infection (Infections and infestations) | 0 (0)
Injection site reaction (General disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (3)
Leukopenia (Investigations) | 13 (41)
Lymphopenia (Investigations) | 9 (20)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy-cranial (Nervous system disorders) | 0 (0)
Neuropathy-motor (Nervous system disorders) | 3 (4)
Neutropenia (Investigations) | 8 (18)
Personality change (Psychiatric disorders) | 1 (1)
Seizure (Nervous system disorders) | 0 (0)
Thrombocytopenia (Investigations) | 2 (2)
Pyramidal tract dysfunction (Nervous system disorders) | 9 (15)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No